CLINICAL TRIAL: NCT01737944
Title: Exposure, Safety and Local Tolerance Study Comparing 3 Routes of Methotrexate (MTX) Administration: Vibex-MTX Device, Subcutaneous (SC)and Intramuscular (IM) in Adult Subjects With Rheumatoid Arthritis
Brief Title: Exposure Study Comparing 3 Routes of Methotrexate (MTX) Administration
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Antares Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MTX-10-001
Record Dates: First submitted 2012-11-27; First posted 2012-11-30 (Estimated); Results first posted 2014-02-25 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-01

CONDITIONS: Rheumatoid Arthritis
Keywords: methotrexate injection, subcutaneous, autoinjector
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 10mg Methotrexate (MTX) Group (Experimental): Treatment Arm A - SC injection with Vibex device, Treatment Arm B - SC injection without device and Treatment Arm C - IM injection
  Interventions: Drug: Methotrexate (MTX)
- 15mg Methotrexate (MTX) Group (Experimental): Treatment Arm A - SC injection with Vibex device, Treatment Arm B - SC injection without device and Treatment Arm C - IM injection
  Interventions: Drug: Methotrexate (MTX)
- 20mg Methotrexate (MTX) Group (Experimental): Treatment Arm A - SC injection with Vibex device, Treatment Arm B - SC injection without device and Treatment Arm C - IM injection
  Interventions: Drug: Methotrexate (MTX)
- 25mg Methotrexate (MTX) Group (Experimental): Treatment Arm A - SC injection with Vibex device, Treatment Arm B - SC injection without device and Treatment Arm C - IM injection
  Interventions: Drug: Methotrexate (MTX)

INTERVENTIONS:
Drug: Methotrexate (MTX) — Vibex MTX Device
  Other Names: Device with MTX

SUMMARY:
Pharmacokinetics (PK) study

DETAILED DESCRIPTION:
To compare the pharmacokinetic (PK) profiles of methotrexate (MTX) following a subcutaneous (SC) injection of MTX using the Vibex device to that obtained after an SC injection of MTX without using the device and to that obtained after an intramuscular (IM) injection of MTX in adult subjects with rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* Male or female >18 years of age with diagnosed Rheumatoid Arthritis(RA).

Exclusion Criteria:

* Chronic or acute renal disease
* Any other clinically significant disease or disorder which, in the opinion of the investigator, might put the subject at risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan J Kivitz, MD;CPI, Principal Investigator — Altoona Center for Clinical Research
Locations (1):
- Altoona Center for Clinical Research, Duncansville, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at 2 sites in the US. Approximately equal number of subjects on 10 mg, 15 mg, 20 mg and 25 mg doses were recruited. The dose group was determined by the Investigator based on subject's current therapeutic regimen of MTX and disease status. The patient's dose was the same for the entire study.
Pre-assignment Details: The order of Methotrexate (MTX) treatment arms (A-SC injection with Vibex-MTX device, B-SC injection without device and C-IM Injection) were randomly assigned and dosing was separated by interval of atleast 7 days to allow for washout before the next treatment was administered.
Groups:
- 10mg MTX Group; 15mg MTX Group; 20mg MTX Group; 25mg MTX Group: [administered via randomized sequence and crossover of Treatment Arm A -SC injection with Vibex MTX device, Treatment Arm B -SC injection without device and Treatment Arm C -IM Injection]
Period: Overall Study
Arm/Group | 10mg MTX Group | 15mg MTX Group | 20mg MTX Group | 25mg MTX Group
Started | 9 | 9 | 9 (10 patients randomized, one patient discontinued before first study drug dose) | 9 (10 patients randomized, one patient discontinued before first study drug dose)
Completed | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 38 subjects were randomized to a treatment sequence. Two subjects discontinued prior to receiving the first study drug dose. Safety Population = 36 subjects who received study drug and completed all study visits. All 36 subjects were included in Pharmacokinetic Population. No discontinuations after first study drug dose.
Groups:
- 10mg MTX Group; 15mg MTX Group; 20mg MTX Group; 25mg MTX Group: [Administered via randomized sequence and crossover of Treatment Arm A, Treatment Arm B and Treatment Arm C]
- Total: Total of all reporting groups
Arm/Group | 10mg MTX Group | 15mg MTX Group | 20mg MTX Group | 25mg MTX Group | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 7 | 7 | 27
  >=65 years | 2 | 3 | 2 | 2 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (10.97) | 63.4 (7.26) | 60.8 (6.18) | 63.0 (6.80) | 62.1 (7.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 6 | 7 | 25
  Male | 2 | 4 | 3 | 2 | 11
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 9 | 9 | 36

OUTCOME MEASURES:

1. Primary Outcome: Bioequivalence Based Upon Dose-Normalized AUC[0-Inf] for MTX
Description: Dose-normalized area under the curve from time zero to infinity (AUC[0-inf]/Dose) for each treatment
Time Frame: 24 Hour period
Population: The Population was defined as all randomized subjects who received at least 1 dose of study drug and who had at least 1 valid post-dose plasma concentration value.
Measure: Mean (Standard Deviation); unit: ng*hr/mL/mg
Groups:
- Treatment Arm A: Subcutaneous (SC) injection with the Vibex MTX device
- Treatment Arm B: SC injection of MTX without the device
- Treatment Arm C: Intramuscular (IM) injection of MTX
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 36 | 36 | 36
ng*hr/mL/mg | 118.14 (42.300) [55.65 to 213.94] | 122.63 (40.648) [80 to 125] | 116.71 (41.394) [80 to 125]
Statistical Analysis 1: Comparison: Treatment Arm A vs Treatment Arm B; Test type: Non-Inferiority or Equivalence — The bioequivalence of Methotrexate following Treatment A - SC injection with the Vibex MTX device and Treatment B - SC injection without the device was established if the 90% CI for the geometric LS Mean ratios of AUC(0-inf)/Dose were within the range of 80% to 125%; Test / Reference Ratio = 96.24, 90% CI 2-sided [92.33 to 100.31]
Statistical Analysis 2: Comparison: Treatment Arm A vs Treatment Arm C; Test type: Non-Inferiority or Equivalence — The bioequivalence of Methotrexate following Treatment A-SC injection with the Vibex MTX device and Treatment C-IM injection was established if the 90% CI for the geometric LS Mean ratios of AUC(0-inf)/Dose were within the range of 80% to 125%; Test / Reference Ratio = 101.28, 90% CI 2-sided [97.17 to 105.56]

2. Primary Outcome: Bioequivalence Based Upon Dose-Normalized AUC[0-24] for MTX
Description: Dose-normalized area under the curve from time zero to 24 hours post-dose (AUC[0-24]/Dose) for each treatment
Time Frame: 24 Hour period
Population: Dose-normalized MTX PK parameter AUC(0-24)/Dose used for comparison
Measure: Mean (Standard Deviation); unit: ng*hr/mL/mg
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 36 | 36 | 36
ng*hr/mL/mg | 116.60 (40.963) | 121.08 (39.405) | 122.63 (40.648)
Statistical Analysis 1: Comparison: Treatment Arm A vs Treatment Arm B; Test type: Non-Inferiority or Equivalence — The bioequivalence of Methotrexate following Treatment A-SC injection with the Vibex MTX device and Treatment B-SC injection was established if the 90% CI for the geometric LS Mean ratios of AUC(0-24)/Dose were within the range of 80% to 125%; Test / Reference Ratio = 96.22, 90% CI 2-sided [92.32 to 100.28]
Statistical Analysis 2: Comparison: Treatment Arm A vs Treatment Arm C; Test type: Non-Inferiority or Equivalence — The bioequivalence of Methotrexate following Treatment A-SC injection with the Vibex MTX device and Treatment C-IM injection was established if the 90% CI for the geometric LS Mean ratios of AUC(0-24)/Dose were within the range of 80% to 125%; Test / Reference Ratio = 101.14, 90% CI 2-sided [97.06 to 105.40]

3. Primary Outcome: Bioequivalence Based Upon Dose-Normalized Cmax for MTX
Description: Dose-normalized maximum observed concentration for each treatment
Time Frame: 24 Hour period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL/mg
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 36 | 36 | 36
ng/mL/mg | 21.43 (8.310) | 22.38 (10.263) | 23.37 (7.188)
Statistical Analysis 1: Comparison: Treatment Arm A vs Treatment Arm B; Test type: Non-Inferiority or Equivalence — The bioequivalence of Methotrexate following Treatment A-SC injection with the Vibex MTX device and Treatment B-SC injection without the device was established if the 90% CI for the geometric LS Mean ratios of Cmax/Dose were within the range of 80% to 125%; Test / Reference Ratio = 96.76, 90% CI 2-sided [87.93 to 106.47]
Statistical Analysis 2: Comparison: Treatment Arm A vs Treatment Arm C; Test type: Non-Inferiority or Equivalence — The bioequivalence of Methotrexate following Treatment A-SC injection with the Vibex MTX device and Treatment C-IM injection was established if the 90% CI for the geometric LS Mean ratios of Cmax/Dose were within the range of 80% to 125%; Test / Reference Ratio = 89.79, 90% CI 2-sided [81.61 to 98.78]

ADVERSE EVENTS:
Time Frame: The Safety Population was defined as all randomized subjects who received at least 1 dose of study drug. The Safety Population included 36 subjects.
Description: Adverse events were classified by treatment at onset. Any adverse event that occurred on Day 1 (after check-in) for a given treatment period was assigned to the treatment for that period.
Groups:
- 10mg MTX; 15mg MTX; 20mg MTX; 25mg MTX: [Administered via randomized sequence and crossover of Treatment A, Treatment B and Treatment C]
Arm/Group | 10mg MTX | 15mg MTX | 20mg MTX | 25mg MTX
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 1/9 | 0/9 | 2/9 | 1/9
OTHER ADVERSE EVENTS (reported when occurring in more than 2.8% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10mg MTX (N=9) | 15mg MTX (N=9) | 20mg MTX (N=9) | 25mg MTX (N=9)
Maculopapular rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — AE Occurred During Treatment A
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — AE Occurred During Treatment A
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — AE Occurred During Treatment B
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — AE Occurred During Treatment B

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less